CLINICAL TRIAL: NCT04887168
Title: An Investigation Into the Effectiveness of Differing Treatment Intensities on a Group-based Psychoeducational Intervention for Complex Interpersonal Trauma Symptomatology With Male Offenders
Brief Title: Survive & Thrive Trial With Male Offenders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Edinburgh Napier University (Other)
Responsible Party: Principal Investigator, Adam Louis Mahoney, Lecturer / Chartered Forensic Psychologist, Edinburgh Napier University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2765584
Record Dates: First submitted 2021-04-28; First posted 2021-05-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Complex Post-Traumatic Stress Disorder
MeSH Terms: interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: non-randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressed (Experimental): Treatment delivered at higher intensity - twice weekly
  Interventions: Behavioral: Survive & Thrive
- Spaced (Experimental): Treatment delivered at lower intensity - once weekly
  Interventions: Behavioral: Survive & Thrive

INTERVENTIONS:
Behavioral: Survive & Thrive — Psychoeducational Intervention: Survive & Thrive (Ferguson, 2008; Mahoney et al, 2018). A total of 10 manualised sessions of approximately 1.5 hour duration are offered. Individual sessions run using an educational format and in an informal setting, with a strong emphasis on avoiding individual disclosures. Groups will be delivered utilising a multi-disciplinary work force consisting of mental health staff in a ratio of 2 per group. Groups will consist of a maximum of 8-10 participants

SUMMARY:
Previous research has concluded that prison populations have particularly high rates of interpersonal trauma. There is however concern that these issues have been largely overlooked and misunderstood in the work undertaken with male offenders. The importance of addressing these concerns can be seen in the greater occurrence of mental health problems and higher reconviction rates often reported by prisoners with histories of interpersonal trauma. This study seeks to investigate complex trauma and associated symptomatology can be effectively ameliorated and whether differences in delivery intensity impact on how interventions respond most effectively to this group of survivors' needs. This is particularly relevant for forensic mental health services located in prisons, which are tasked with the care and rehabilitation of large populations of survivors.

DETAILED DESCRIPTION:
Central to this study will be the use of non-randomised control design whereby all participants will receive treatment at the trial sites they are currently located at. The sites will deliver the intervention at different intensities either weekly (ie 'spaced') or twice weekly ('compressed'). As such the trial design is a pragmatic response to the resources made available to facilitate this trial. A sample of n = 196 male prisoners with a history of complex interpersonal trauma will be drawn from the 2 participating UK prison establishments. Participants will be initially identified by routine 'generic' and mental health assessments that consider a range of social, health and offending behaviour related needs. Those prisoners whose prior assessments indicate a history of childhood or adulthood trauma will be invited to participate in a one-off interview. Information during interviews will be collected by means of standardised questionnaires regarding the nature and extent of lifetime traumatic events and current psychopathology.

All trial participants will continue their usual psychological, psychiatric, and medical care during the study. Data collection interviews will be carried out in designated interview areas within the prison or any other suitable place of their choosing. All interviews will be conducted by a research assistant, who will have experience in working with adults with complex trauma and mental health concerns.

Psychoeducational Intervention: Survive & Thrive (S&T). The 'present focussed' group format is designed to be part of the process of stabilisation of clients presenting difficulties prior to embarking on work with the traumatic elements of their experiences. Survive & Thrive was designed to help clients achieve stabilisation in a resource efficient way, while at the same time providing service users with support while they are on waiting lists to access further treatment. The focus of this intervention is therefore primarily on ensuring safety, stabilisation and affect management skills.

A total of 10 manualised sessions of approximately 1.5 hour duration are offered. Individual sessions run using an educational format and in an informal setting, with a strong emphasis on avoiding individual disclosures. Groups will be delivered utilising a multi-disciplinary work force consisting of mental health staff in a ratio of 2 per group. Groups will consist of a maximum of 8-10 participants per group and whilst they will be randomly selected in accordance with the procedure outlined about a local treatment manager (psychology manager) will ensure that issues all security concerns and group dynamics that might potentially mitigate the effectiveness of the intervention are accounted for. All professionals who facilitate the delivery of the programme will have a background in applied psychology or mental health and will have received standardised three-day training on the delivery of the intervention and an additional day to account for the adjustments made to S&T to assist with delivery in this population and setting. Regular supervision will also be provided during the delivery of the programme.

Inclusion Criteria: All convicted male inmates over the age of 18 years old at the trial sites who indicate a history of interpersonal complex trauma will be invited to participate in this study. It should be noted that potential participants may present with different clusters of PTSD and CPTSD symptoms.

A completer and an intention to treat analysis will be performed. Irrespective of time of termination all participants will be invited for an end point blind assessment. Premature termination due to recovery will be at any time, whilst patients terminating prematurely due to lack of improvement must complete at least 7 sessions in the study before they can be classified as completers. A maximum of 10 sessions will be offered as part of the project. Qualitative and quantitative procedures will analyse resultant data to establish acceptability of the intervention and the treatment efficacy of differing treatment intensities.

ELIGIBILITY:
Inclusion Criteria:

All convicted male inmates over the age of 18 years old who indicate a history of interpersonal complex trauma will be invited to participate in this study. The ITQ will be used to identify the presence of complex trauma. It should be noted that potential participants may present with different clusters of PTSD and CPTSD symptoms; it is thought that this should not compromise the overall integrity of the study (Facer-Irwin et al, 2021). The selection process should also help to ensure:

* An adequate level of mental and physical health and substance misuse stability so as to enable them to cope with the requirements of the intervention as determined by the local Multi-disciplinary Mental Health Team (MDMHT).
* Willing to participate for therapeutic and rehabilitative reasons and to have voluntarily given their written consent.
* Serving a sentence of 6-months or more and able to complete all follow up assessments prior to their liberation.
* Have a sufficient level of literacy skills that will enable them to engage with the course written material. Learning disabilities or difficulties will be considered on a case by case basis as discussed with the Treatment Manager.
* Located in a mainstream residential location.

Exclusion Criteria:

It is intended that as fewer prisoners as possible will be excluded from this study. Therefore, the following exclusion criteria are primarily based on ensuring the safety or the individual, other participants/staff and the good order and functioning of the prison establishment. This should include;

* Prisoners who present as a high risk of institutional violence and requiring segregation from mainstream residential units
* Those who are on frequent observations for suicide and self-harm at any time in the week prior to the intervention starting.
* Enemies and those who have formed intimate relationships with each other whilst in custody will also be allocated to separate groups to ensure appropriate therapeutic dynamics. This will be undertaken in consultation with staff from establishment security department.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 196 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire about Process of Recovery | Week 0 (T1: 'Pre'), Week 5 (T2: 'Post'), Week 10 (T3: 'FU1') Week 15 (T4: 'FU2') , Week 20 (T5: 'FU3')
  Measures change on self-reported improvements in mental health and general wellbeing. This 22-item measure is developed from service users' accounts of recovery and seeks to elicit responses about aspects of recovery that are meaningful to participants. Each item is scored on a 4-point scale, from 0 ('disagree strongly') to 4 ('agree strongly') with higher scores are indicative of recovery.

SECONDARY OUTCOMES:
General Anxiety Disorder-7 | Week 0 (T1: 'Pre'), Week 5 (T2: 'Post'), Week 10 (T3: 'FU1') Week 15 (T4: 'FU2') , Week 20 (T5: 'FU3')
  Measures change on self reported anxiety symptomatology. This 7-item instrument is used to briefly measure and screen for general anxiety general anxiety symptoms across various settings and populations. Items are measured on a 3 point scale from 0 ('not at all') to 3 ('nearly every day'). Symptom amelioration is indicated in a reduction in total scores.
Patient Health Questionnaire-9 | Week 0 (T1: 'Pre'), Week 5 (T2: 'Post'), Week 10 (T3: 'FU1') Week 15 (T4: 'FU2') , Week 20 (T5: 'FU3')
  Measures change on symptomatology associated with depressive disorders. Items are measured on a 3-point scale from 0 ('not at all') to 3 ('nearly every day'). Symptom amelioration is indicated in a reduction in total scores.
Clinical Outcome in Routine Evaluation -10 | Week 0 (T1: 'Pre'), Week 5 (T2: 'Post'), Week 10 (T3: 'FU1') Week 15 (T4: 'FU2') , Week 20 (T5: 'FU3')
  Measures change in self reported psychological distress to track overall progress during the course of treatment. Items are measured on a 4-point scale from 0 ('not at all') to 4 ('most or all of the time'). Symptom amelioration is indicated in a reduction in total scores.
PTSD Checklist for DSM 5 | Week 0 (T1: 'Pre'), Week 5 (T2: 'Post'), Week 10 (T3: 'FU1') Week 15 (T4: 'FU2') , Week 20 (T5: 'FU3')
  Measures change on PTSD symptomatology between time points. Participants respond on a 5-point scale, ranging from 'not at all' to 'extremely' as to how much the specific symptom was a problem for them over the past month. Scores are calculated resulting in a total severity score from 0 to 80. A reduction in scores indicating symptom improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Hakanpaa, PhD, Study Director — Edinburgh Napier University

IPD SHARING:
Plan to Share IPD: No